CLINICAL TRIAL: NCT01493791
Title: Evaluation of Whether the Selective Progesterone Receptor Modulator CDB-2914 Can Reduce Bleeding in Premenopausal Women With Abnormal Uterine Bleeding: A Pilot Study
Brief Title: CDB-2914 for Abnormal Uterine Bleeding in Premenopausal Women
Status: Withdrawn | Phase: Early Phase 1 | Type: Interventional
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Parallel | Purpose: Treatment
Other Study IDs: 120015; 12-CH-0015
Record Dates: First submitted 2011-12-15; First posted 2011-12-16 (Estimated); Last update posted 2019-12-17 (Actual); Status verified 2013-07-24

CONDITIONS: Urogenital Abnormalities
Keywords: CDB-2914; Abnormal Urine Bleeding; Abnormal Uterine Bleeding
MeSH Terms: conditions — Urogenital Abnormalities; Metrorrhagia | interventions — ulipristal

INTERVENTIONS:
Drug: CDB-2914

SUMMARY:
Background:

- CDB-2914 is a hormone that blocks progesterone, which is necessary for maintaining pregnancy. In women with fibroid tumors, CDB-2914 shrank the tumors. In many cases, menstrual periods stopped during treatment. Because CDB-2914 decreased or stopped menstrual bleeding in women with fibroids, it may be able to treat abnormal periods in women without fibroids.

Objectives:

- To see whether CDB-2914 can treat abnormal uterine bleeding in premenopausal women.

Eligibility:

- Premenopausal women who have abnormal uterine bleeding that is not caused by fibroids.

Design:

* Participants will be screened with a physical exam and medical history. They will also have blood and urine tests. An ultrasound with fluid of the uterus will test for fibroids. Uterine cells will be collected for biopsy.
* For the next three menstrual cycles, participants will take either CDB-2914 or a placebo. Treatment will be studied with blood tests and symptom diaries.
* At the end of the treatment, participants have three options. They can have surgery at the Clinical Center or have another 3 months of CDB-2914. The third option is to stop treatment at the Clinical Center.
* Surgery will be either uterine ablation or hysterectomy. Only women older than age 33 may have a hysterectomy. Blood and urine samples will be collected after surgery.
* Both surgery and further treatment participants will have followup exams.
* All participants will have a final followup exam 1 year after stopping treatment....

DETAILED DESCRIPTION:
Abnormal uterine bleeding is the most common gynecologic complaint in reproductive aged women. Medical treatment of abnormal uterine bleeding has high failure rates and surgical management remains the primary, definitive therapy. Most women undergoing hysterectomy for abnormal bleeding failed a therapeutic trial of medical management. Consequently, development of an efficacious, new medical treatment for abnormal uterine bleeding is urgently needed. Many of these reproductive aged women also need contraception. Ulipristal acetate (UPA), a novel progesterone receptor modulator developed at the NIH, has promise as an effective medical treatment for abnormal uterine bleeding and as a contraceptive agent. In women with symptomatic fibroids, UPA significantly reduced fibroid size, stopped menstrual bleeding and led to an increase in red blood cell hemoglobin. It also inhibited release of an egg from the ovaries (ovulation) without reducing estrogen levels or causing hot flashes, making contraception a potential future use.

This study will evaluate UPA effects on estrogen production and ovulation, and will determine whether it reduces bleeding in women who have abnormal uterine bleeding as assessed by the Menorrhagia Impact Questionnaire (MIQ) and menstrual calendars. Women with an anatomic abnormality of the uterus are not eligible to participate. Participants will take UPA (10 mg daily by mouth) or a similar-appearing inactive pill (placebo) for approximately 90 days. Women will be randomly assigned to receive daily UPA 10 mg, or a daily placebo tablet, during the initial three-month period. The participants and the investigators will not be informed of the treatment group. To understand the effects of UPA on the uterus and its lining (endometrium), women will have studies before and at the end of UPA treatment, including ultrasound imaging of the uterus after injection of a small amount of sterile saline into the uterine cavity, and a biopsy of the endometrium to examine the tissue under the microscope. Before and while taking study agent, women will record daily bleeding and complete the MIQ monthly. During the treatment period, blood will be taken weekly to measure hormone levels (to evaluate ovulation blockage), and monthly to evaluate safety. At the end of the randomized study period, the research team will offer participants additional options of UPA or surgical therapy. Women may choose surgical therapy at the NIH or may elect other treatment options elsewhere.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Female gender - to evaluate effects in the target population for clinical trials
* History of abnormal uterine bleeding documented by menorrhagia impact questionnaire (MIQ) and menstrual calendar
* Anovulatory and ovulatory women will be included
* In good health. Chronic medication use is acceptable except for glucocorticoid use. Other chronic medication use may be acceptable at the discretion of the research team. Interval use of over-the counter drugs is acceptable but must be recorded.
* Ovulatory women will be defined as those who have menstrual cycles of 24 35 days and a progesterone value > 3.0 pg/mL between 5 and 9 days after in-home documentation of an LH surge
* Anovulatory women will be defined as those without an in-house LH surge in whom progesterone values 3 and 4 weeks after menses are < 3.0 ng/mL
* Hemoglobin > 10 g/dL (for those wishing surgery); iron may be administered to improve red blood cell counts
* Willing and able to comply with study requirements
* Age 25-40
* Using mechanical (condoms, diaphragms), sterilization or abstinence methods of contraception for the duration of the study
* Negative urine pregnancy test
* BMI less than or equal to 33, if a surgical candidate or less than or equal to 35, if not a surgical candidate.
* Creatinine less than 1.3 mg/dL
* Liver function tests within 130 percent of upper limit
* Women who elect surgery must state that they do not desire further fertility.
* Endometrial biopsy without endometrial hyperplasia or neoplasia
* Normal cervical cytology screening within the last 12 months

EXCLUSION CRITERIA:

* Significant abnormalities in the history, physical or laboratory examination
* Pregnancy
* Lactation
* Use of oral, injectable or inhaled glucocorticoids or megesterol within the last year
* History of malignancy within the past 5 years
* Vaginal Bleeding in context of anatomic abnormality, endometrial neoplasia or hyperplasia, cervical, vaginal, or vulvar neoplaisa or preneoplastic pathology
* Use of estrogen or progesterone-containing compounds, such as oral contraceptives and hormone replacement therapy, within 8 weeks of study entry, including transdermal, injectable, vaginal and oral preparations
* Current use of agents known to induce hepatic P450 enzymes; use of imidazoles
* Current use of GnRH analogs or other compounds that affect menstrual cyclicity
* Use of herbal medication having estrogenic or antiestrogenic effects within the past 3 months
* FSH > 20 IU/mL
* Untreated cervical dysplasia
* Need for interval use of narcotics
* Abnormal adnexal/ovarian mass
* Contradiction to anesthesia, for women planning surgery
* Leiomyomata, polyps or other anatomic causes of vaginal bleeding
* Previous participation in the study
* Thrombocytopenia defined as platelets < 150,000
* Patients with known abnormal breast pathology

Ages: 25 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2011-11-08; Primary Completion 2013-07-24 (Actual); Study Completion 2013-07-24 (Actual)

PRIMARY OUTCOMES:
Primary outcome parameters will include bleeding symptoms evaluated by Menorrhagia Impact Questionnaire (MIQ), composite bleeding score, endometrial hyperplasia, changes in hemoglobin (g/dL)

SECONDARY OUTCOMES:
Quality of life as measured by surveys.

CONTACTS AND LOCATIONS:
Overall Officials: Alicia Y Christy, M.D., Principal Investigator — Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD)

REFERENCES:
- [Background] Batista MC, Cartledge TP, Zellmer AW, Merino MJ, Axiotis C, Loriaux DL, Nieman LK. Delayed endometrial maturation induced by daily administration of the antiprogestin RU 486: a potential new contraceptive strategy. Am J Obstet Gynecol. 1992 Jul;167(1):60-5. doi: 10.1016/s0002-9378(11)91627-5. PMID 1442957
- [Background] Bushnell DM, Martin ML, Moore KA, Richter HE, Rubin A, Patrick DL. Menorrhagia Impact Questionnaire: assessing the influence of heavy menstrual bleeding on quality of life. Curr Med Res Opin. 2010 Dec;26(12):2745-55. doi: 10.1185/03007995.2010.532200. Epub 2010 Nov 3. PMID 21043553
- [Background] Cadepond F, Ulmann A, Baulieu EE. RU486 (mifepristone): mechanisms of action and clinical uses. Annu Rev Med. 1997;48:129-56. doi: 10.1146/annurev.med.48.1.129. PMID 9046951